CLINICAL TRIAL: NCT00640276
Title: A Prospective Comparative Clinical Study to Identify Efficacy and Safety of Pitavastatin in Patients With a Metabolic Syndrome
Brief Title: Safety and Efficacy Study of Pitavastatin in Patient With a Metabolic Syndrome
Acronym: ProPit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP_PTV_706
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Hypercholesterolemia; Metabolic Syndrome
Keywords: pitavastatin; metabolic syndrome; metabolic syndrome risk score; hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Metabolic Syndrome | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T (Active Comparator): Lifestyle modification + active drug(Pitavastatin)
  Interventions: Drug: pitavastatin
- C (Other): Lifestyle Modification
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Drug: pitavastatin — Pitavastatin 2mg daily once
  Other Names: Livaro
  Arms: T
Behavioral: Lifestyle Modification — conducting mainly exercises and diet
  Arms: C

SUMMARY:
We will identify the influence of long-term treatment of Pitavastatin compared to non-treatment control group on the metabolic syndrome by evaluation of a change of metabolic syndrome component score. And we will additionally observe the changes of CVD risk factors like lipid profile, abdominal fat, insulin resistance and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75
* Patients with LDL ≥ 100mg/dL
* Patients with metabolic syndrome

  1. IFG: Fasting glucose ≥ 100mg/dL
  2. Abdominal Obesity: Waist circumference: men≥90cm,women≥85cm
  3. 1 or more of the following

     1. Triglyceride ≥ 150mg/dL
     2. HDL-C: men < 40mg/dL, women < 50mg/dL
     3. Blood pressure: SBP ≥ 130mmHg or DBP ≥ 85mmHg or subject receiving anti-hypertensive treatment

Exclusion Criteria:

* uncontrolled hypertension (DBP ≥ 95mmHg)
* taking diabetic drugs or with HbA1c > 8%
* LDL ≥ 190mg/dL or Triglyceride ≥ 400mg/dL
* coronary heart disease or other diseases caused by artherosclerosis
* malignancy within 6 months
* Serum creatinine ≥ 2.0mg/dL
* ALT or AST ≥ ULN*2.5
* CPK ≥ ULN*2
* hypothyroidism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
A change of metabolic syndrome risk component | 48week

SECONDARY OUTCOMES:
Changes of cardiometabolic profiles : lipid profiles, hs-CRP, adiponectin, HMW adiponectin | 48week
Changes of abdominal visceral fat | 48week
Changes of insulin resistance : OGTT(75g), HOMA | 48week

CONTACTS AND LOCATIONS:
Overall Officials: Chang Beom Lee, Study Chair — Hanyang Univ. Guri Hospital; Hak Chul Jang, Study Chair — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Bundang-gu, Gyeonggi-do
  - Hanyang Univ. Guri Hospital, Guri-si, Gyeonggi-do